CLINICAL TRIAL: NCT01658670
Title: HEART Camp: Promoting Adherence to Exercise in Patients With Heart Failure
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Wayne State University (Other); Henry Ford Health System (Other); University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0608-11-FB; 1R01HL112979 (NIH)
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: Heart failure; exercise; adherence; quality of life
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) exercise group (Active Comparator): The EUC group is provided paid access to the exercise facility and has access to regular facility staff for the 18 month study period.
  Interventions: Behavioral: Enhanced Usual Care Group
- HEART Camp (HC) Intervention group (Experimental): The HC intervention group will be provided paid access to the exercise facility for the 18 month study period and will also receive the cognitive-behavioral intervention (knowledge, attitudes, self-efficacy, behavioral self-management skills and social support) delivered using both group-based and individual-based strategies.
  Interventions: Behavioral: HEART Camp (HC) Intervention Group

INTERVENTIONS:
Behavioral: Enhanced Usual Care Group — The EUC group is provided access to the exercise facility and regular facility staff for the 18 month study period.
  Arms: Enhanced Usual Care (EUC) exercise group
Behavioral: HEART Camp (HC) Intervention Group — The HC intervention group will be provided access to the exercise facility for the 18 month study period and will also receive the cognitive-behavioral intervention (knowledge, attitudes, self-efficacy, behavioral self-management skills and social support) delivered using both group-based and individual-based strategies.
  Arms: HEART Camp (HC) Intervention group

SUMMARY:
The purpose of this study is to determine the efficacy of the Heart Failure Exercise and Resistance Training (HEART) Camp behavioral exercise training intervention on long-term adherence to exercise at 18 months in patients with heart failure. The central hypothesis is that the HEART Camp intervention group (HC) will have significantly better adherence to exercise at 18 months.

DETAILED DESCRIPTION:
The objective of this prospective randomized two-group repeated measures experimental design is to determine the efficacy of the HEART (Heart Failure Exercise and Resistance Training) Camp behavioral exercise training intervention on long-term adherence to exercise at 18 months in patients with HF. A sample size of 246 subjects with heart failure will be recruited over a 3 year period. All subjects will receive a cardiopulmonary exercise test and 9 supervised exercise training sessions during a 3 week run-in period prior to randomization. Subjects completing 6 of 9 training sessions will be randomized to the HEART Camp Intervention group (HC) or to an enhanced usual care (EUC) exercise group. The HC intervention group will receive cognitive-behavioral strategies that address the intervention components of knowledge, attitudes, self-efficacy, behavioral self-management skills and social support. The EUC group is provided access to the exercise facility and regular facility staff for the 18 month study period. Our central hypothesis is that the HC group will have significantly better adherence to exercise at 18 months. We will test our hypothesis with the following Specific Aims: Aim 1. To evaluate the effect of HEART Camp on adherence to exercise (measured by self-report and validated by heart rate monitor); Aim 2. To evaluate which components of the HEART Camp intervention mediate the effects of the intervention on adherence; Aim 3. To evaluate the effect of HEART Camp on specific health outcomes; Aim 4. To explore selected demographic variables (age, race, gender, body mass index and left ventricular ejection fraction) as potential moderators of the effect of the HEART Camp intervention on adherence; and Aim 5. To explore the perceptions and experiences that contextualize exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure (stage C chronic HF confirmed by echocardiography and clinical evaluation)
* 19 years of age or greater
* able to speak and read English
* telephone access in home
* Stable pharmacologic therapy per guidelines for past 30 days

Exclusion Criteria:

* clinical evidence of decompensated HF
* unstable angina pectoris
* myocardial infarction, coronary artery bypass surgery, or biventricular pacemaker within the past 6 weeks
* orthopedic or neuromuscular disorders preventing participation in aerobic exercise and strength/resistance training
* participation in 3 times per week aerobic exercise during the past 8 weeks
* cardiopulmonary stress test results that preclude safe exercise training
* plans to move more than 50 miles from the exercise site within the next year
* peak oxygen uptake (pVO2) in women>21mL kg min and in men >24mLkg min
* planned or current pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Adherence to exercise. | 18 months
  Adherence to exercise with 18 months as the primary outcome time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bunny J Pozehl, PhD, RN, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Nebraska Medical Center, College of Nursing, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pozehl BJ, Duncan K, Hertzog M, McGuire R, Norman JF, Artinian NT, Keteyian SJ. Study of adherence to exercise in heart failure: the HEART camp trial protocol. BMC Cardiovasc Disord. 2014 Nov 29;14:172. doi: 10.1186/1471-2261-14-172. PMID 25433674
- [Result] Pozehl BJ, McGuire R, Duncan K, Kupzyk K, Norman J, Artinian NT, Deka P, Krueger SK, Saval MA, Keteyian SJ. Effects of the HEART Camp Trial on Adherence to Exercise in Patients With Heart Failure. J Card Fail. 2018 Oct;24(10):654-660. doi: 10.1016/j.cardfail.2018.06.007. Epub 2018 Aug 16. PMID 30010027
- [Result] Pozehl BJ, Mcguire R, Duncan K, Hertzog M, Deka P, Norman J, Artinian NT, Saval MA, Keteyian SJ. Accelerometer-Measured Daily Activity Levels and Related Factors in Patients With Heart Failure. J Cardiovasc Nurs. 2018 Jul/Aug;33(4):329-335. doi: 10.1097/JCN.0000000000000464. PMID 29538050
- [Result] Brawner CA, Ehrman JK, Myers J, Chase P, Vainshelboim B, Farha S, Saval MA, McGuire R, Pozehl B, Keteyian SJ. Exercise Oscillatory Ventilation: Interreviewer Agreement and a Novel Determination. Med Sci Sports Exerc. 2018 Feb;50(2):369-374. doi: 10.1249/MSS.0000000000001423. PMID 28902683
- [Derived] Salahshurian E, Pozehl BJ, Lundgren SW, Bills S, Pandey A, Carbone S, Alonso WW. 'Working me to life': longitudinal perceptions from adults with heart failure with preserved ejection fraction enrolled in an exercise training clinical trial. Eur J Cardiovasc Nurs. 2024 Oct 21;23(7):763-770. doi: 10.1093/eurjcn/zvae049. PMID 38597735
- [Derived] Alonso WW, Kupzyk KA, Norman JF, Lundgren SW, Fisher A, Lindsey ML, Keteyian SJ, Pozehl BJ. The HEART Camp Exercise Intervention Improves Exercise Adherence, Physical Function, and Patient-Reported Outcomes in Adults With Preserved Ejection Fraction Heart Failure. J Card Fail. 2022 Mar;28(3):431-442. doi: 10.1016/j.cardfail.2021.09.003. Epub 2021 Sep 15. PMID 34534664